CLINICAL TRIAL: NCT04230798
Title: Effect of an Injury Prevention Program on the Lower Limb Stability in Young Volleyball
Brief Title: Effect of an Injury Prevention Program on the Lower Limb Stability in Young Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Mario Albaladejo-Saura, Master´s Degree, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Injury prevention volleyball
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Sports Injury
Keywords: Sport; Strength; Plyometrics; Core stability; Prevention program; Young athletes
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group did not perform any specific exercise program nor injury prevention program. They continued their normal training routine
- Prevention program (Experimental): This group performed two sessions per week of the injury prevention program. The program included strength training, plyometrics and core stability training.
  Interventions: Other: Injury prevention program

INTERVENTIONS:
Other: Injury prevention program — The intervention program consisted in 16 sessions, performed during eight weeks, twice per week. Intervention group performed 20 minutes sessions before their habitual volleyball training. The structure of the prevention program consisted in a warm up, a lower limb strength exercise; two core exercises; a lower limb plyometric exercise, and a lower limb stability exercise. While the injury prevention program was being performed, both groups continued with their volleyball training sessions.
  Arms: Prevention program

SUMMARY:
Volleyball players have a high injury risk as a consequence of the specific sport characteristics, as repetitive jumps and falls. The aim of the present study was to evaluate the effects of a multidisciplinary injury prevention program on lower limb stability in young volleyball players. It was spected to improve the stability of the lowe limb and, as a consecuence, to reduce the injury risk of the most common injuries in volleyball.

DETAILED DESCRIPTION:
A sample of 29 players were included in this study. The experimental group was formed by 18 players, while the control group was formed by 11 players. Sample characteristics for both groups are shown in Table 1. The inclusion criteria for the sample selection were: 1) to be aged between 14 and 18 years old; 2) to train in volleyball twice or three times a week, for at least an hour and a half per session; 3) to take part in federated competitions regularly; 4) to have been competing in volleyball for at least two seasons. The exclusion criteria were: 1) to leave the training or the competition during the study; 2) to suffer an injury at the beginning of the intervention program or during its implementation; 3) to miss more than 25% of the training sessions during the intervention program. Lastly, three players from the experimental group were excluded from the statistical analysis because they interrupted their volleyball practice.

The study was approved for the institutional ethics committee. An explanatory letter was given to the participants and their parents and an informed consent form was signed by the parents of the participants.

The intervention program consisted of 16 sessions, performed for eight weeks, twice per week. The intervention group performed 20-minute sessions before their habitual volleyball training. The structure of the prevention program consisted in a warm up, a lower limb strength exercise; two core exercises; a lower limb plyometric exercise, and a lower limb stability exercise. While the injury prevention program was being performed, both groups continued with their regular volleyball training sessions. The sessions designed for each day can be observed in Figure 1.

Strength training was oriented to increase the strength-endurance capacity of the players. It was focused on the quadriceps, hamstrings, gluteus maximus and gluteus medius, spinal erectors, transverse abdominal, obliques and rectus abdominis. These muscles perform flexion and extension of the knee and the hip, and stabilize the spine, hip and knee. A range of 10-20 repetitions were performed of each exercise, or 15-30 seconds in the case of isometric exercises. Plyometric training was focused on the lower limbs. A total volume of 40 jumps and landings were performed in each session, so volume was controlled by the number of jumps performed according to the guidelines published by the National Strength Conditioning Association (NSCA). Stability training was divided into three groups depending on if they were performed without equipment, with a volleyball ball, or after a landing.

Two measurements were carried out. The first one, a week before the intervention (pre-test) and, the second one a week after the 8 weeks of the injury prevention program (post-test). The participants answered a questionnaire about previous sport injuries of the lower limbs in the pre-test. A laterality test was performed to confirm the dominant side of the subjects. After that, some anthropometric variables and stability with a force platform and the Y-Balance test were taken randomly.

Height was evaluated with a stadiometer (SECA, Germany) and weight with a scale SECA 862 (SECA, Germany) in the pre-test. Iliospinale height was measured with a segmometer (Cescorf, Brazil) in the pre- and post-test. These measurements were taken according to the Society for the Advancement of Kinanthropometry (ISAK) protocols, and completed by a level 3 ISAK kinanthropometrist, twice or three times if there was a difference between the first two measurements greater than 1%. The final value was the mean or median depending on the number of measurements taken, two or three, respectively.

Stability with a force platform was measured using a MuscleLab force plate (Ergotest Innovation S.A., Norway). The tests consisted on a frontal jump from a distance of 40% of the subject´s height, and a lateral jump from a distance of 33% of the subject´s height. Players had to land in the force platform in a one-leg stance and hold the position for ten seconds. There was an obstacle between the jumping zone and the force platform that was 30 cm in height for the frontal jump and 15 cm for the lateral jump. Players were told to perform the jump without any restrictions in arm movement, but they had to place them on their hips when they landed on the platform, while staring towards the front. The jump was valid if they were able to maintain the position during the established time without touching the platform with the other foot or losing balance. To minimize the risk of error, the participants jumped from a wooden platform located at the same height with respect to the ground as the force platform, built ad hoc. They performed frontal or lateral jumps and dominant or non-dominant leg landings in a random order. Subjects rested three minutes between attempts. Each participant made two valid frontal jumps and two valid lateral jumps. The better of the two attempts was included in the statistical analyses. The five seconds after the first contact of the subjects on the platform were collected. To relativize the data obtained from the force platform, the following formula was used: [√ (0-FX) 2- (0-FY) 2+ (body weight-FZ) 2] / body weight, with FX being the center of the pressure sway in the mid-lateral axis (X axis), and FY the center of the pressure sway in the front-rear axis (Y axis), and FZ the vertical reaction force (Z axis).

The Y-Balance test consisted of a three-axis version (anterior, post-lateral and post-medial) of the Star Excursion Balance test. The validated instrument Y-Balance Test Kit (FMS, U.S.A.) was used to register the data. The subjects performed the test barefoot. While on a single leg stance, the subject was asked to reach the maximum distance with the free limb in the anterior, posteromedial, and posterolateral directions in relation to the standing foot. The instructions given to the participants were to keep the toes behind the line in the platform, and push the reach indicator without stepping in any direction with the free limb. The test order started with the anterior direction, followed by posteromedial and posterolateral directions. They had to place their hands on their hips during the test. If all of these instructions were followed, the attempt would be valid. Three non-consecutive trials were performed by each player, where the stance leg for the first trial was randomized. Subjects rested for three minutes between attempts. The testing protocol was designed based on previous publications. The best of three attempts for each direction and leg were collected for the statistical analyses. The test results were relativized with the player's iliospinale height. The following fórmula was used: [(anterior axis value+posteromedial axis value+posterolateral axis value)/(3 x iliospinale height)] x 100.

All the tests were performed by expert researchers who were already familiar with the measurement tests. Both measurements, pre-test and post-test, were recorded by the same blinded researcher for each test and performed under the same measurement conditions, in the same room and at a standard temperature of 25°C. The players should not have performed any type of physical exercise prior to the measurements, nor strenuous physical exercise in the 24 hours prior to the data collection.

Descriptive statistical analyses was performed for all the variables. The mean and standard deviation were calculated for the quantitative variables and frequency and percentage for the categorical variables. The Shapiro-Wilks test was used to determine the distribution of the sample and the Levene's test to determine the homogeneity of variances. Following a normal data distribution, the statistical analysis was performed based on parametric tests. The differences in the characteristics of the sample between groups were analyzed with a t-test for independent samples. To analyze whether the effects of the prevention program were significant, a two-factor MANOVA analysis (group and measurement) was performed, thus studying the effect on the dependent variables (stability) exerted by intra-subject (measurement) and inter-subject (group). A post hoc Bonferroni adjustment was selected to determine the interactions between pairs. Statistical significance was established at a value of p <0.05. The SPSS program (version 23.0, IBM, USA) was used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* to train volleyball twice or three times a week, at least an hour and half each session
* to take part in federated competitions regularly
* to have been competing in volleyball at least two seasons

Exclusion Criteria:

* to leave the training or the competition during the study
* to suffer an injury at the beginning of the intervention program or during the process
* to miss more than 25% of the training during the intervention program

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Dynamic stability change | Change of Dynamic stability after 8 weeks
  Dynamic stability was assesed whith the Y-Balance test device and protocol
Static stability change | Change of Static stability after 8 weeks
  Assesed with a forces platform. After a frontal jump and lateral jump respectively

SECONDARY OUTCOMES:
Height change | Change of heigth after 8 weeks
  Height measured in centimetres with a stadiometer
Weight change | Change of weight after 8 weeks
  Body mass assesment
Leg length change | Change of the leg length after 8 weeks
  Length measured from the trochanterion to the floor
Sport and record of previous injuries | At the begining of the study
  Interview with a questionnaire designed ad hoc

CONTACTS AND LOCATIONS:
Overall Officials: Mario Albaladejo-Saura, Master, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No